CLINICAL TRIAL: NCT03817229
Title: Fostering Medication Adherence in Children With Epilepsy Using mHealth Technology
Brief Title: Epilepsy Adherence in Children and Technology (eACT)
Acronym: eACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Medical University of South Carolina (Other); Children's Hospital of Orange County (Other); University of Cincinnati (Other); Nationwide Children's Hospital (Other); North Carolina State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FP00001781; R01NR017794-01A1 (NIH)
Record Dates: First submitted 2018-12-27; First posted 2019-01-25 (Actual); Results first posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-09

CONDITIONS: Epilepsy
Keywords: adherence; mHealth; eHealth; children; caregivers; compliance
MeSH Terms: conditions — Epilepsy; Patient Compliance

STUDY DESIGN:
Intervention Model Description: This a 2-stage, sequential, multiple assignment, randomized trial (SMART) . In Stage 1 (three months long), non-adherent caregivers (< 95%) will be randomized to a mHealth education module and automated digital reminders (control) or the mHealth education module, automated digital reminders, and individualized adherence feedback based on real-time adherence monitoring (treatment) to address the primary barrier of forgetting. At the beginning of Stage 2 (two months long), caregivers randomized to treatment who do not achieve adherence > 95% (response) by the end of Stage 1 will be re-randomized to either continued individualized adherence feedback or individualized adherence feedback augmented with three mHealth problem-solving modules (translated from the PIs existing RCTs) with a therapist.
Who Masked: Care Provider, Investigator
Masking Description: The PI will not be notified of group status or details of participants. The healthcare provider will also not know which group participants are randomized to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Active Comparator): mHealth education module and automated digital reminders
  Interventions: Behavioral: Education microlearning sessions; Behavioral: Automated digital reminders
- Treatment Group-Individualized Feedback Only (Experimental): mHealth education module, automated digital reminders, and individualized adherence feedback.
  Interventions: Behavioral: Education microlearning sessions; Behavioral: Automated digital reminders; Behavioral: Individualized Adherence Feedback Report
- Treatment Group-Individualized Feedback + Problem-Solving (Experimental): mHealth education module, automated digital reminders, individualized adherence feedback, and 2 problem solving sessions with a therapist.
  Interventions: Behavioral: Education microlearning sessions; Behavioral: Automated digital reminders; Behavioral: Problem-solving mHealth module; Behavioral: Individualized Adherence Feedback Report

INTERVENTIONS:
Behavioral: Education microlearning sessions — mHealth education microlearning sessions
Behavioral: Automated digital reminders — reminders from electronic monitors based on texts or lights/chimes
Behavioral: Problem-solving mHealth module — mhealht problem solving module with 2 telehealth sessions with a therapist
  Arms: Treatment Group-Individualized Feedback + Problem-Solving
Behavioral: Individualized Adherence Feedback Report — Individual Adherence Feedback reports sent to parents weekly
  Arms: Treatment Group-Individualized Feedback + Problem-Solving; Treatment Group-Individualized Feedback Only

SUMMARY:
Fifty-eight percent of children with new-onset epilepsy do not take their antiepileptic drugs (AEDs) as prescribed, which is associated with continued seizures, mortality, poor quality of life, and high healthcare costs. Evidence-based adherence interventions are lacking and critically needed, especially for children with epilepsy, who represent an underserved population in pediatrics. The current proposal is a mHealth sequential, multiple assignment, randomized trial (SMART) focused on providing education, automated digital reminders, and individualized adherence feedback, as well as teaching problem-solving skills, with the goal of improving adherence and quality of life and decreasing seizures and health care utilization.

DETAILED DESCRIPTION:
Non-adherence to antiepileptic drugs (AEDs) is a common problem (i.e., 58% of patients have some level of non-adherence) for young children with newly diagnosed epilepsy, with potentially devastating consequences. AED non-adherence is associated with a 3-fold increased risk of seizures, poor quality of life, inaccurate clinical decision-making, and higher health care utilization and costs. One of the primary barriers to adherence is forgetting, which may be particularly amenable to mHealth (mobile technology in healthcare) interventions. Despite the critical need to develop and implement interventions to improve adherence, there are few family-based interventions for young children with epilepsy and their families. One existing intervention is highly promising; however, this intervention requires six in-person sessions, which can be impossible for families who lack routine access to tertiary specialty care due to time, financial, or transportation constraints. Thus, unmet medical and psychosocial needs of the underserved pediatric epilepsy population are perpetuated and compounded by limited access to this state of the art care. The overall goal is to test a mHealth adherence intervention that is easily accessible using a stepped up care model based on individual needs. This stepped up care model will conserve patient, family, and provider time, costs and resources. The aim of this multi-site R01 is to conduct a two-stage, sequential, multiple assignment, randomized trial (SMART) to evaluate the effectiveness of mHealth intervention strategies for improving AED adherence in caregivers of young children with epilepsy. A two-month baseline period will be followed by two stages. In Stage 1 (3-months long), non-adherent caregivers (< 95%) will be randomized to a mHealth education module and automated digital reminders (control) or the mHealth education module, automated digital reminders, and individualized adherence feedback based on real-time adherence monitoring (treatment) to address the primary barrier of forgetting. At the beginning of Stage 2 (two months long), caregivers randomized to treatment who do not achieve adherence > 95% (response) by the end of Stage 1 will be re-randomized to either continued individualized adherence feedback or individualized adherence feedback augmented with two mHealth problem-solving modules (translated from the PIs existing RCTs) with a therapist. Thus, there are three intervention strategies embedded in this SMART: #1 control, #2 treatment, and #3 problem-solving augmented treatment if nonresponsive at three months. The primary outcome is electronically-monitored adherence and secondary outcomes include seizure severity/frequency, quality of life, and healthcare utilization. If the aims of the project are achieved, this study would have a large impact on pediatric epilepsy, with the potential to change clinical practice for treating non-adherence. The SMART design would allow the investigators to identify patients who are most likely to respond to interventions and step up care with more time- and resource-intensive interventions (i.e., problem-solving with a therapist via the web), when necessary.

ELIGIBILITY:
Inclusion criteria:

1. Children ages 2-12 years
2. Epilepsy diagnosis < 2 years
3. Ability to read/speak English

Exclusion criteria:

1. Major comorbid neurodevelopmental or medical disorders (e.g., Autism, diabetes)
2. Plan to wean AEDs for 18 months

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 268 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Avani Modi, Ph.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (4):
- United States (4):
  - Childrens Hospital of Orange County, Orange, California
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
Prior to sharing, all data will be de-identified in a HIPAA-compliant fashion. Data sets will be carefully reviewed to make sure that information such as age and gender cannot be used to gather additional information that could potentially identify individual subjects. All modalities of data will be shared, including raw and aggregate data. Descriptors for all variables shared will be included to prevent misuse or confusion. Any analytical methods utilized to assess the data will be defined in shared formats. In addition, treatment manuals related to problem-solving and mHealth modules will also be shared after completion of the trial for future use.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 12 months after completion of the study
Access Criteria: Requested from the PI

REFERENCES:
- [Derived] Wagner JL, Patel AD, Huszti H, Schmidt M, Smith G, Bhatia S, Guilfoyle SM, Lang A, Buschhaus S, Williams S, Ardo J, Davidian M, Modi AC. The eACT study design and methods: A sequential, multiple assignment, randomized trial of A novel adherence intervention for youth with epilepsy. Contemp Clin Trials. 2024 Dec;147:107739. doi: 10.1016/j.cct.2024.107739. Epub 2024 Nov 10. PMID 39532238

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from four sites: Cincinnati Children's Hospital Medical Center, Medical University of South Carolina, Children's Hospital of Orange County, and Nationwide Children's Hospital. Participants were recruited through epilepsy clinics from April 2019-September 2023.
Pre-assignment Details: Following recruitment, participants were in a run-in period of 2 months. All participants who demonstrated adherence > 95% ended study participation at the end of the 2-month run-in period and were ineligible for randomization.
Groups:
- Treatment Group (E+ADR+IAF in Stage 1 and remained in Stage 2): mHealth education module, automated digital reminders, and individualized adherence feedback (stage 1 SMART). After three months of intervention, the treatment group will be evaluated for responsiveness (> 95%) based on the 30-day adherence outcome (stage 2 SMART). These were participants in the treatment group demonstrate adherence > 95%, and continued with the treatment arm of receiving automated digital reminders and individualized adherence feedback.
  Education microlearning sessions: mHealth education microlearning sessions
  Automated digital reminders: reminders from electronic monitors based on texts or lights/chimes
  Individualized Adherence Feedback Report: Individual Adherence Feedback reports sent to parents weekly
- Treatment Group (E+ADR+IAF) non-responsive but continue IAF: mHealth education module, automated digital reminders, and individualized adherence feedback (stage 1 SMART). After three months of intervention, the treatment group will be evaluated for responsiveness (> 95%) based on the 30-day adherence outcome (stage 2 SMART). These participants were considered non-responsive (adherence </= 95%) after Stage one and re-randomized to continued automated digital reminders and individualized adherence feedback.
  Education microlearning sessions: mHealth education microlearning sessions
  Automated digital reminders: reminders from electronic monitors based on texts or lights/chimes
  Individualized Adherence Feedback Report: Individual Adherence Feedback reports sent to parents weekly
- Treatment Group (E+ADR+IAF+PS) non-responsive and PS added: mHealth education module, automated digital reminders, and individualized adherence feedback (stage 1 SMART). After three months of intervention, the treatment group will be evaluated for responsiveness (> 95%) based on the 30-day adherence outcome (stage 2 SMART). These participants were considered non-responsive (adherence </= 95%) after Stage one and re-randomized to two additional problem-solving sessions with a telehealth therapist.
  Education microlearning sessions: mHealth education microlearning sessions
  Automated digital reminders: reminders from electronic monitors based on texts or lights/chimes
  Problem-solving sessions with a therapist via telehealth: Two sessions over two months.
Period: Intervention Period-Stage 1
Arm/Group | Control Group | Treatment Group (E+ADR+IAF in Stage 1 and remained in Stage 2) | Treatment Group (E+ADR+IAF) non-responsive but continue IAF | Treatment Group (E+ADR+IAF+PS) non-responsive and PS added
Started | 89 | 179 | 0 (Had not reached Stage 2 yet) | 0
Completed | 83 | 167 | 0 (Had not reached Stage 2 yet) | 0
Not Completed | 6 | 12 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 8 | 0 | 0
Not completed — Withdrawn by Study Team | 0 | 1 | 0 | 0
Not completed — Weaned from medication | 0 | 3 | 0 | 0
Period: Intervention Period-Stage 2
Arm/Group | Control Group | Treatment Group (E+ADR+IAF in Stage 1 and remained in Stage 2) | Treatment Group (E+ADR+IAF) non-responsive but continue IAF | Treatment Group (E+ADR+IAF+PS) non-responsive and PS added
Started | 83 | 48 (Participants were re-randomized after Stage 1 into two groups) | 56 (Participants were re-randomized after Stage 1 into two groups) | 63 (Participants were re-randomized after Stage 1 into two groups)
Completed | 82 | 48 | 55 | 49
Not Completed | 1 | 0 | 1 | 14
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 10
Not completed — Withdrawal by Study Team | 0 | 0 | 0 | 3
Not completed — Weaned from medication | 0 | 0 | 0 | 1
Period: Post-Intervention
Arm/Group | Control Group | Treatment Group (E+ADR+IAF in Stage 1 and remained in Stage 2) | Treatment Group (E+ADR+IAF) non-responsive but continue IAF | Treatment Group (E+ADR+IAF+PS) non-responsive and PS added
Started | 82 | 48 | 55 | 49
Completed | 69 | 47 | 49 | 42
Not Completed | 13 | 1 | 6 | 7
Not completed — Withdrawal by Subject | 6 | 0 | 2 | 2
Not completed — Withdrawal by Study Team | 3 | 1 | 1 | 4
Not completed — Weaned from medication | 3 | 0 | 2 | 1
Not completed — Transferred care to another institution | 1 | 0 | 0 | 0
Not completed — Change in parental guardianship | 0 | 0 | 1 | 0
Period: Follow-up 1
Arm/Group | Control Group | Treatment Group (E+ADR+IAF in Stage 1 and remained in Stage 2) | Treatment Group (E+ADR+IAF) non-responsive but continue IAF | Treatment Group (E+ADR+IAF+PS) non-responsive and PS added
Started | 69 | 47 | 49 | 42
Completed | 54 | 36 | 45 | 38
Not Completed | 15 | 11 | 4 | 4
Not completed — Ineligible for this follow-up visit due to study timing | 7 | 4 | 4 | 3
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 0
Not completed — Withdrawal by Study Team | 3 | 1 | 0 | 0
Not completed — Wean from medication | 3 | 4 | 0 | 1
Not completed — Transferred care to another hospital | 1 | 0 | 0 | 0
Period: Follow-up 2
Arm/Group | Control Group | Treatment Group (E+ADR+IAF in Stage 1 and remained in Stage 2) | Treatment Group (E+ADR+IAF) non-responsive but continue IAF | Treatment Group (E+ADR+IAF+PS) non-responsive and PS added
Started | 54 | 36 | 45 | 38
Completed | 45 | 33 | 41 | 33
Not Completed | 9 | 3 | 4 | 5
Not completed — Ineligible for this follow-up visit due to study timing | 4 | 3 | 1 | 4
Not completed — Withdrawal by Subject | 2 | 0 | 1 | 1
Not completed — Withdrawal by Study Team | 2 | 0 | 1 | 0
Not completed — Wean from medication | 1 | 0 | 0 | 0
Not completed — Transferred care | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Group: mHealth education module, automated digital reminders, and individualized adherence feedback (stage 1 SMART). After three months of intervention, the treatment group will be evaluated for responsiveness (> 95%) based on the 30-day adherence outcome (stage 2 SMART). If participants in the treatment group demonstrate adherence > 95%, they will continue with the treatment arm of receiving automated digital reminders and individualized adherence feedback. If they are deemed to be non-responsive (adherence < 95%), they will be re-randomized to either: 1) continued automated digital reminders and individualized adherence feedback or 2) a mHealth problem solving module with three therapist-guided problem-solving sessions.
  Education microlearning sessions: mHealth education microlearning sessions
  Automated digital reminders: reminders from electronic monitors based on texts or lights/chimes
  Problem-solving mHealth module: mhealht problem solving module with 2 telehealth sessions with a therapist
  Individualized Adherence Feedback Report: Individual Adherence Feedback reports sent to parents weekly
- Total: Total of all reporting groups
Arm/Group | Control Group | Treatment Group | Total
Number analyzed (Participants) | 89 | 179 | 268
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.4 (3.1) | 7.4 (3.0) | 7.4 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 96 | 140
  Male | 45 | 83 | 128
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 35 | 51
  Not Hispanic or Latino | 73 | 144 | 217
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 1 | 11 | 12
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 8 | 23 | 31
  White | 69 | 116 | 185
  More than one race | 8 | 17 | 25
  Unknown or Not Reported | 1 | 10 | 11
Region of Enrollment [Number; unit: participants]
  United States | 89 | 179 | 268

OUTCOME MEASURES:

1. Primary Outcome: Anti-seizure Medication Adherence Rate
Description: Electronically monitored adherence, as measured by the Simplemed+ pillboxes or Adheretech bottles will be used as the primary outcome to calculate an adherence rate. A monthly adherence rate for antiseizure medication is calculated for Month 5, which ranges from 0-100%, with higher scores reflecting higher adherence.
Time Frame: Stage 1 (Month 5)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Treatment Group (E+ADR+IAF): mHealth education module, automated digital reminders, and individualized adherence feedback (stage 1 SMART). After three months of intervention, the treatment group will be evaluated for responsiveness (> 95%) based on the 30-day adherence outcome (stage 2 SMART).
  Education microlearning sessions: mHealth education microlearning sessions
  Automated digital reminders: reminders from electronic monitors based on texts or lights/chimes
  Individualized Adherence Feedback Report: Individual Adherence Feedback reports sent to parents weekly
Arm/Group | Control Group | Treatment Group (E+ADR+IAF)
Number analyzed (Participants) | 83 | 167
score on a scale | 68.93 (35.65) | 77.23 (27.29)

2. Secondary Outcome: Antiseizure Medication Adherence Rate
Description: lectronically monitored adherence, as measured by the Simplemed+ pillboxes or Adheretech bottles will be used as the primary outcome to calculate an adherence rate. A monthly adherence rate for antiseizure medication is calculated for Month 8, which ranges from 0-100%, with higher scores reflecting higher adherence.
Time Frame: Month 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Treatment Group (E+ADR+IAF in Stage 1 and remained in Stage 2) | Treatment Group (E+ADR+IAF) non-responsive but continue IAF | Treatment Group (E+ADR+IAF+PS) non-responsive and PS added
Number analyzed (Participants) | 70 | 47 | 51 | 43
score on a scale | 58.80 (32.29) | 74.42 (32.02) | 48.87 (33.27) | 54.76 (34.98)

3. Secondary Outcome: Antiseizure Medication Adherence Rate
Description: lectronically monitored adherence, as measured by the Simplemed+ pillboxes or Adheretech bottles will be used as the primary outcome to calculate an adherence rate. A monthly adherence rate for antiseizure medication is calculated for Month 7, which ranges from 0-100%, with higher scores reflecting higher adherence.
Time Frame: Month 7 (Stage 2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Treatment Group (E+ADR+IAF in Stage 1 and remained in Stage 2) | Treatment Group (E+ADR+IAF) non-responsive but continue IAF | Treatment Group (E+ADR+IAF+PS) non-responsive and PS added
Number analyzed (Participants) | 73 | 48 | 54 | 46
score on a scale | 71.68 (31.99) | 91.66 (14.98) | 68.52 (25.93) | 79.71 (23.05)

4. Secondary Outcome: Global Assessment of Severity of Epilepsy
Description: The GASE is a item measure, ranging from 1-7, with 7 representing worse seizure severity. GASE was dichotomized with a 0 or 1 rating. Participants who received a GASE severity score of 1 or 2 were given a 0 score and those who received a GASE score of 3-7 were given a 1 score. In this context, a GASE category of 0 is the lower severity rating.
Time Frame: Months 8-13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Treatment Group (E+ADR+IAF in Stage 1 and remained in Stage 2) | Treatment Group (E+ADR+IAF) non-responsive but continue IAF | Treatment Group (E+ADR+IAF+PS) non-responsive and PS added
Number analyzed (Participants) | 75 | 44 | 52 | 46
units on a scale | 0.28 (0.45) | 0.25 (0.44) | 0.33 (0.47) | 0.24 (0.43)

5. Secondary Outcome: PedsQL Epilepsy Module-Impact (Parent Report)
Description: The Pediatric Quality of Life (PedsQL) Epilepsy Module is a 29-item epilepsy-specific HRQOL measure for youth with epilepsy between the ages of 2 and 18 years with excellent reliability and validity. A total of five different subscales comprise this measure, including Cognitive, Impact, Sleep, Executive Functioning, and Mood/Behavior. Parallel and developmentally appropriate forms exist for both youth and their caregiver, who record their answers using a 5-point Likert scale ranging from 0 = never a problem to 4 = almost always a problem. Scores range from 0-100, with higher scores representing better HRQOL. Internal consistency for the subscales range from 0.70 to 0.94.
Time Frame: Month 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Treatment Group (E+ADR+IAF in Stage 1 and remained in Stage 2) | Treatment Group (E+ADR+IAF) non-responsive but continue IAF | Treatment Group (E+ADR+IAF+PS) non-responsive and PS added
Number analyzed (Participants) | 65 | 45 | 40 | 40
score on a scale | 78.76 (18.25) | 81.67 (18.52) | 81.01 (21.57) | 85.07 (16.52)

6. Secondary Outcome: Seizure Severity Adapted for Children Scale-Total Score
Description: Seizure Severity Scale Adapted for Children is a measure of seizure severity via parent-report. This caregiver questionnaire is nine-items assessing the child's seizure severity. Items focus on the intrusiveness, frequency, length, and disruptiveness of seizures. Items are scored from 0-3 and a mean is calculated across items for a Total score. Higher scores reflect greater seizure severity.
Time Frame: Month 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Treatment Group (E+ADR+IAF in Stage 1 and remained in Stage 2) | Treatment Group (E+ADR+IAF) non-responsive but continue IAF | Treatment Group (E+ADR+IAF+PS) non-responsive and PS added
Number analyzed (Participants) | 66 | 44 | 42 | 41
score on a scale | 0.92 (0.46) | 0.91 (0.58) | 0.92 (0.66) | 0.86 (0.60)

7. Secondary Outcome: Seizure Freedom
Description: Seizure Freedom is a dichotomous variable regarding the absence or presence of seizures over a 4 month period of time. Participants were given a score of 0 if they had no seizures and a score of 1 if they had any seizures during that time frame. Thus, a score of 0 represents seizure freedom while a score of 1 represents the presence of seizures.
Time Frame: Months 8-11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Treatment Group (E+ADR+IAF in Stage 1 and remained in Stage 2) | Treatment Group (E+ADR+IAF) non-responsive but continue IAF | Treatment Group (E+ADR+IAF+PS) non-responsive and PS added
Number analyzed (Participants) | 71 | 48 | 50 | 48
units on a scale | 0.54 (0.50) | 0.50 (0.51) | 0.60 (0.49) | 0.58 (0.50)

8. Secondary Outcome: Antiseizure Medication Adherence Rate
Description: lectronically monitored adherence, as measured by the Simplemed+ pillboxes or Adheretech bottles will be used as the primary outcome to calculate an adherence rate. A monthly adherence rate for antiseizure medication is calculated for Month 14, which ranges from 0-100%, with higher scores reflecting higher adherence.
Time Frame: Month 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Treatment Group (E+ADR+IAF in Stage 1 and remained in Stage 2) | Treatment Group (E+ADR+IAF) non-responsive but continue IAF | Treatment Group (E+ADR+IAF+PS) non-responsive and PS added
Number analyzed (Participants) | 44 | 35 | 33 | 27
score on a scale | 50.26 (33.46) | 72.76 (36.16) | 43.26 (31.72) | 59.02 (31.00)

9. Secondary Outcome: Global Assessment of Severity of Epilepsy
Description: as for outcome 4
Time Frame: Months 14-19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Treatment Group (E+ADR+IAF in Stage 1 and remained in Stage 2) | Treatment Group (E+ADR+IAF) non-responsive but continue IAF | Treatment Group (E+ADR+IAF+PS) non-responsive and PS added
Number analyzed (Participants) | 53 | 33 | 40 | 34
units on a scale | 0.19 (0.39) | 0.18 (0.39) | 0.35 (0.48) | 0.35 (0.49)

10. Secondary Outcome: PedsQL Epilepsy Module-Impact (Parent Report)
Description: as for outcome 5
Time Frame: Month 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Treatment Group (E+ADR+IAF in Stage 1 and remained in Stage 2) | Treatment Group (E+ADR+IAF) non-responsive but continue IAF | Treatment Group (E+ADR+IAF+PS) non-responsive and PS added
Number analyzed (Participants) | 34 | 29 | 34 | 30
score on a scale | 82.2 (16.64) | 82.14 (19.76) | 82.03 (21.82) | 85.19 (14.11)

11. Secondary Outcome: PedsQL Epilepsy Module-Cognition (Parent Report)
Description: as for outcome 5
Time Frame: Month 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Treatment Group (E+ADR+IAF in Stage 1 and remained in Stage 2) | Treatment Group (E+ADR+IAF) non-responsive but continue IAF | Treatment Group (E+ADR+IAF+PS) non-responsive and PS added
Number analyzed (Participants) | 65 | 45 | 40 | 40
score on a scale | 62.15 (27.43) | 68.89 (27.74) | 63.56 (28.51) | 64.35 (29.68)

12. Secondary Outcome: PedsQL Epilepsy Module-Cognition (Parent Report)
Description: as for outcome 5
Time Frame: Month 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Treatment Group (E+ADR+IAF in Stage 1 and remained in Stage 2) | Treatment Group (E+ADR+IAF) non-responsive but continue IAF | Treatment Group (E+ADR+IAF+PS) non-responsive and PS added
Number analyzed (Participants) | 34 | 29 | 34 | 30
score on a scale | 61.90 (27.11) | 69.20 (25.97) | 63.85 (26.66) | 65.03 (30.09)

13. Secondary Outcome: PedsQL Epilepsy Module-Sleep (Parent Report)
Description: as for outcome 5
Time Frame: Month 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Treatment Group (E+ADR+IAF in Stage 1 and remained in Stage 2) | Treatment Group (E+ADR+IAF) non-responsive but continue IAF | Treatment Group (E+ADR+IAF+PS) non-responsive and PS added
Number analyzed (Participants) | 65 | 45 | 40 | 40
score on a scale | 51.92 (25.74) | 59.07 (23.78) | 59.27 (23.56) | 62.71 (23.64)

14. Secondary Outcome: PedsQL Epilepsy Module-Sleep (Parent Report)
Description: as for outcome 5
Time Frame: Month 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Treatment Group (E+ADR+IAF in Stage 1 and remained in Stage 2) | Treatment Group (E+ADR+IAF) non-responsive but continue IAF | Treatment Group (E+ADR+IAF+PS) non-responsive and PS added
Number analyzed (Participants) | 34 | 29 | 34 | 30
score on a scale | 54.53 (23.44) | 57.76 (27.09) | 62.01 (22.49) | 61.53 (27.28)

15. Secondary Outcome: PedsQL Epilepsy Module-Executive Functioning (Parent Report)
Description: as for outcome 5
Time Frame: Month 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Treatment Group (E+ADR+IAF in Stage 1 and remained in Stage 2) | Treatment Group (E+ADR+IAF) non-responsive but continue IAF | Treatment Group (E+ADR+IAF+PS) non-responsive and PS added
Number analyzed (Participants) | 65 | 45 | 40 | 40
score on a scale | 51.70 (28.51) | 63.80 (24.43) | 56.46 (30.40) | 59.43 (28.58)

16. Secondary Outcome: PedsQL Epilepsy Module-Executive Functioning (Parent Report)
Description: as for outcome 5
Time Frame: Month 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Treatment Group (E+ADR+IAF in Stage 1 and remained in Stage 2) | Treatment Group (E+ADR+IAF) non-responsive but continue IAF | Treatment Group (E+ADR+IAF+PS) non-responsive and PS added
Number analyzed (Participants) | 34 | 29 | 34 | 30
score on a scale | 55.27 (32.87) | 59.05 (27.56) | 58.54 (27.98) | 57.71 (29.69)

17. Secondary Outcome: PedsQL Epilepsy Module-Mood/Behavior (Parent Report)
Description: as for outcome 5
Time Frame: Month 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Treatment Group (E+ADR+IAF in Stage 1 and remained in Stage 2) | Treatment Group (E+ADR+IAF) non-responsive but continue IAF | Treatment Group (E+ADR+IAF+PS) non-responsive and PS added
Number analyzed (Participants) | 34 | 29 | 34 | 30
score on a scale | 61.91 (20.67) | 70.00 (18.37) | 64.56 (19.12) | 68.50 (24.88)

18. Secondary Outcome: PedsQL Epilepsy Module-Mood/Behavior (Parent Report)
Description: as for outcome 5
Time Frame: Month 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Treatment Group (E+ADR+IAF in Stage 1 and remained in Stage 2) | Treatment Group (E+ADR+IAF) non-responsive but continue IAF | Treatment Group (E+ADR+IAF+PS) non-responsive and PS added
Number analyzed (Participants) | 65 | 45 | 40 | 40
score on a scale | 63.08 (21.61) | 74.44 (17.56) | 69.62 (19.13) | 69.12 (22.64)

19. Secondary Outcome: Seizure Freedom
Description: as for outcome 7
Time Frame: Month 14-17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Treatment Group (E+ADR+IAF in Stage 1 and remained in Stage 2) | Treatment Group (E+ADR+IAF) non-responsive but continue IAF | Treatment Group (E+ADR+IAF+PS) non-responsive and PS added
Number analyzed (Participants) | 48 | 39 | 40 | 36
units on a scale | 0.69 (0.47) | 0.64 (0.49) | 0.55 (0.50) | 0.64 (0.49)

20. Secondary Outcome: Seizure Severity Adapted for Children Scale-Total Score
Description: as for outcome 6
Time Frame: Month 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Treatment Group (E+ADR+IAF in Stage 1 and remained in Stage 2) | Treatment Group (E+ADR+IAF) non-responsive but continue IAF | Treatment Group (E+ADR+IAF+PS) non-responsive and PS added
Number analyzed (Participants) | 35 | 31 | 35 | 29
score on a scale | 0.84 (0.52) | 0.87 (0.50) | 0.81 (0.63) | 0.64 (0.52)

21. Secondary Outcome: Emergency Room and Urgent Care Visits Combined
Description: Emergency Room and Urgent Care Visits Combined (Healthcare utilization) - Number of emergency room visits based on medical chart review and caregiver report. Higher scores reflect more visits.
Time Frame: Months 8-14
Measure: Mean (Standard Deviation); unit: number of emergency room visits
Arm/Group | Control Group | Treatment Group (E+ADR+IAF in Stage 1 and remained in Stage 2) | Treatment Group (E+ADR+IAF) non-responsive but continue IAF | Treatment Group (E+ADR+IAF+PS) non-responsive and PS added
Number analyzed (Participants) | 55 | 41 | 43 | 37
number of emergency room visits | 0.33 (0.84) | 0.12 (0.40) | 0.28 (0.55) | 0.32 (0.63)

22. Secondary Outcome: Hospitalizations (Healthcare Utilization)
Description: Number of inpatient hospitalization based on medical chart review and caregiver report. Higher numbers mean a higher level of inpatient hospitalizations.
Time Frame: Months 8-14
Measure: Mean (Standard Deviation); unit: number of inpatient hospitalizations
Arm/Group | Control Group | Treatment Group (E+ADR+IAF in Stage 1 and remained in Stage 2) | Treatment Group (E+ADR+IAF) non-responsive but continue IAF | Treatment Group (E+ADR+IAF+PS) non-responsive and PS added
Number analyzed (Participants) | 55 | 41 | 43 | 37
number of inpatient hospitalizations | 0.13 (0.47) | 0.17 (0.38) | 0.30 (0.47) | 0.32 (0.63)

ADVERSE EVENTS:
Time Frame: 20 months
Description: The Stage 1 non-responsive group is divided into two groups in Stage 2: 1) Treatment Group (E+ADR+IAF) Non-responsive But Continue IAF and 2) Treatment Group (E+ADR+IAF+PS) Non-responsive and PS Added. Thus, we did not present the combined Stage 1 data as they are reported separately and would redundant. n=12 participants withdrew from the study during Stage 1 treatment and thus were excluded from these data.
Arm/Group | Control Group | Treatment Group (E+ADR+IAF in Stage 1 and remained in Stage 2) | Treatment Group (E+ADR+IAF) non-responsive but continue IAF | Treatment Group (E+ADR+IAF+PS) non-responsive and PS added
All-Cause Mortality (participants affected / at risk) | 0/89 | 0/48 | 0/56 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/89 | 0/48 | 1/56 | 0/63
Other Adverse Events (participants affected / at risk) | 35/89 | 13/48 | 24/56 | 21/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=89) | Treatment Group (E+ADR+IAF in Stage 1 and remained in Stage 2) (N=48) | Treatment Group (E+ADR+IAF) non-responsive but continue IAF (N=56) | Treatment Group (E+ADR+IAF+PS) non-responsive and PS added (N=63)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=89) | Treatment Group (E+ADR+IAF in Stage 1 and remained in Stage 2) (N=48) | Treatment Group (E+ADR+IAF) non-responsive but continue IAF (N=56) | Treatment Group (E+ADR+IAF+PS) non-responsive and PS added (N=63)
Medical complications not related to epilepsy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Medical complications not related to epilepsy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Medical complications not related to epilepsy (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Medical complications not related to epilepsy (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Medical complications not related to epilepsy (General disorders) | 2 (6) | 0 (0) | 0 (0) | 0 (0)
Medical complications not related to epilepsy (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Medical complications not related to epilepsy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical complications not related to epilepsy (Infections and infestations) | 13 (18) | 3 (3) | 6 (8) | 7 (19)
Medical complications not related to epilepsy (Injury, poisoning and procedural complications) | 7 (8) | 0 (0) | 5 (5) | 3 (3)
Medical complications not related to epilepsy (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Medical complications not related to epilepsy (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical complications not related to epilepsy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Medical complications not related to epilepsy (Skin and subcutaneous tissue disorders) | 3 (7) | 0 (0) | 0 (0) | 0 (0)
Medical complications not related to epilepsy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Planned Inpatient/Outpatient Procedures Not Related to Epilepsy (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Planned Inpatient/Outpatient Procedures Not Related to Epilepsy (Surgical and medical procedures) | 1 (1) | 2 (2) | 7 (7) | 2 (2)
Medical complications related to epilepsy (Nervous system disorders) | 9 (24) | 2 (3) | 6 (6) | 7 (9)
Planned Inpatient/Outpatient Procedures Related to Epilepsy (Surgical and medical procedures) | 5 (7) | 3 (4) | 8 (10) | 4 (5)
Psychological Complications (Psychiatric disorders) | 3 (3) | 2 (2) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Health utilization data were not analyzed as the trial took place during the COVID-19 pandemic which affected the comfort of participants going to their emergency room departments and/or inpatient hospitalizations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-03-08): https://cdn.clinicaltrials.gov/large-docs/29/NCT03817229/Prot_001.pdf
  • Statistical Analysis Plan (2025-05-20): https://cdn.clinicaltrials.gov/large-docs/29/NCT03817229/SAP_002.pdf
  • Informed Consent Form (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/29/NCT03817229/ICF_000.pdf